CLINICAL TRIAL: NCT06741345
Title: A Phase 1 Multiple Ascending Dose and Food Effect Trial of BIO 300 Oral Suspension in Healthy Volunteers
Brief Title: Phase 1 BIO 300 Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CL0111-01; W911SR-23-9-0018 (Other Grant/Funding Number: JPEO-CBRND)
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteer Study
Keywords: healthy volunteer; BIO 300 Oral Suspension; Genistein; acute radiation syndrome; radiation; radioprotection; pharmacokinetics; pharmacodynamics; multiple ascending dose; food effect; safety; medical countermeasure
MeSH Terms: conditions — Acute Radiation Syndrome

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose study will enroll three cohorts sequentially. An optional fourth cohort may be enrolled. The food effect study follows a randomized, balanced, single-dose, two-treatment (i.e., fed versus fasted), two-period, crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Multiple Ascending Dose (Experimental): The multiple ascending dose study has a single arm. Three cohorts are enrolled sequentially and given ascending doses of study intervention.
  Interventions: Drug: BIO 300 Oral Suspension
- Food Effect: Fed-Fasted Arm (Experimental): Food effect study arm that is administered the study intervention first under fed conditions and then under fasted conditions following crossover.
  Interventions: Drug: BIO 300 Oral Suspension
- Food Effect: Fasted-Fed (Experimental): Food effect study arm that is administered the study intervention first under fasted conditions and then under fed conditions following crossover.
  Interventions: Drug: BIO 300 Oral Suspension

INTERVENTIONS:
Drug: BIO 300 Oral Suspension — Suspension of genistein nanoparticles for oral administration
  Other Names: genistein nanosuspension

SUMMARY:
This is a two-part study of BIO 300 Oral Suspension in healthy male and female volunteers. The first part is a multiple ascending dose (MAD) study to test the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of the drug when given as daily doses over 14 days. The study will enroll three cohorts each receiving a different daily dose: 2000 mg, 3000 mg, or 4000 mg. A fourth group may be added depending on results on the first three cohorts. Each cohort will include 10 participants (5 men, 5 women), with at least 8 completing all study steps. Participants will follow a special diet low in soy-based foods and will fast before certain doses. Blood samples and health checks will be done throughout the study to assess safety, drug is absorption and distribution in the body (PK), and its effects (PD). Safety will be reviewed after each group finishes to decide if the next dose level is safe to proceed.

The second part of the study is a food effect study to examine how food effects the PK of a single dose of BIO 300 Oral Suspension. This study will enroll 16 participants (8 men, 8 women) and will be split into two groups: one group will take the drug after fasting for 10 hours and the other will take the drug after eating a high-fat meal. After a 7-day break, participants will switch conditions (the previously fasted group will take the drug with food, and the previously fed group will take the drug after fasting). Blood samples and health checks will measure how food influences drug absorption (PK) and safety. Both the MAD study and food effect study aim to ensure the drug is safe and provide data on how it behaves in the body under different conditions.

DETAILED DESCRIPTION:
Part 1: Multiple Ascending Dose Study (MAD): Open-label, ascending dose given once daily for 14 days in healthy volunteers. The study will enroll 3 cohorts (dose levels) sequentially, each with 10 participants (5F/5M) per cohort, so that a minimum of 8 study participants (4F/4M) per cohort complete all study procedures. Participants will follow a diet low in soy isoflavones for 7 days before, during and 7 days after treatment and will be required to fast at least 10 hours before the first, sixth and last dose. BIO 300 Oral Suspension will be administered starting on day 1. The first cohort, Cohort 1, will be administered BIO 300 Oral Suspension at 2000 mg/day once daily for 14 days. If dose escalation criteria are met, Cohort 2 will be administered 3000 mg/day, and similarly if dose escalation criteria are met following Cohort 2, then Cohort 3 will be administered 4000 mg/day. Following the completion of Cohort 3, there will be an option to enroll a fourth cohort at a higher or lower dose depending on the outcomes of the first three cohorts. Participants will be administered BIO 300 Oral Suspension daily during their scheduled clinic visits. Participants will remain in the clinic 12 hours after the first dose, sixth dose and last dose and for observations and blood sample collection for clinical lab assessment, pharmacokinetics (PK) and pharmacodynamics (PD). On the day 1, 6 and 14, participants will remain fasted after dosing for 4 hours until provided a standardized low soy meal after the 4 hour blood draw and after the 8 hour blood draw. Blood sampling and/or observations will be performed on dosing days 1-14 as described in the schedule of events. Participants will return to the clinic on days 15, 16 and 21 after their final dose for blood sampling and/or observations as detailed in the schedule of events. Safety data will be reviewed after the completion of each cohort to approve dose escalation. At the conclusion of all three cohorts, all data will be analyzed to assess safety, PK and PD. If the optional fourth cohort is enrolled, all data (safety, PK and PD) from the fourth cohort will be analyzed at the conclusion of the cohort.

Part 2: Food Effect Study: Following the MAD study, an open-label, single-dose food effect study in healthy volunteers will be conducted. The study will enroll 16 participants (8F/8M), so that a minimum of 12 study participants (6F/6M) complete all study procedures. Study participants will be randomized 1:1 into two cohorts. Cohort 1 will be administered a single BIO 300 Oral Suspension dose under fasted conditions and Cohort 2 will be administered a single BIO 300 Oral Suspension dose under fed conditions. After a 7 day washout period, participants in cohort 1 will receive another dose of BIO 300 Oral Suspension under fed conditions and participants in cohort 2 will receive another dose of BIO 300 Oral Suspension under fasted conditions (cross over design). All participants will follow a diet low in soy isoflavones for 7 days before dosing, during the washout period and for 7 days after dosing. The planned BIO 300 Oral Suspension dose used in this study will be 3000 mg, however this is subject to change following safety and PK data review following the completion of the MAD study above. For fasted dosing, participants will be required to fast for at least 10 hours prior to dosing and for 4 hours after dosing. For fed dosing, participants will receive an FDA-approved high-fat meal with no substitutions (800-1000 calories; approximately 50% of calories derived from fat) following an overnight fast of at least 10 hours. The entire meal will be consumed within 30 minutes, dosing will begin 30 minutes after starting the meal, and participants will fast for 4 hours after dosing. All participants will remain in the clinic 12 hours after each dose for observations and blood sample collection for clinical lab assessment, and PK. All participants will remain fasted (fasted cohort) or fast (fed cohort) after dosing for 4 hours until provided a standardized low soy meal after the 4 hour blood draw and after the 8 hour blood draw. Participants will return to the clinic on day 2 and 3 after dosing for blood sampling and/or observations as detailed in the schedule of events (day 10 and 11 after the second dose). At the conclusion of the study, data will be analyzed from both cohorts to determine safety and PK.

ELIGIBILITY:
INCLUSION: In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Healthy adult, 18-64 years old.
2. BMI 18-30 kg/m2
3. No ingestion of prescription or over-the-counter medications (including dietary and herbal supplements) for 7 days prior to first dose of study drug and no planned use during study participation. Acetaminophen of up to 3 g/day and ibuprofen up to 1 g/day will be allowed at discretion of the Investigator.
4. At the discretion of the Investigator, blood routine, liver and kidney functions are within the controllable range.

   1. Adequate hepatic function as evidenced by ALT, AST or LDH < 1.25X ULN and bilirubin < 1.5X ULN for the reference lab.
   2. Adequate renal function as evidenced by a serum creatinine ≤ 1.5 X ULN for the reference laboratory OR a calculated creatinine clearance of ≥ 60 mL/min by the estimated glomerular filtration rate (eGFR).
   3. Adequate hematopoietic function as evidenced by white blood cells ≥ 3x109 / L and platelets ≥ 100x109 / L.
5. Female study participants must have a negative pregnancy test within 72 hours of the start of treatment.
6. Study participants must agree to abstain from heterosexual intercourse or use an effective method of contraception for 7 days after their last dose. Study participants using hormonal contraception are required to utilize double barrier contraception method for 7 days after their last dose.
7. No nicotine use for 30 days prior to first dose, confirmed by negative cotinine test on day 1.
8. Study participant must agree to abstain from THC use from screening to day 1 and for the duration of the study and agree to abstain from alcohol starting 48 hours prior to day 1 and for the duration of the study.
9. Ability to read and provide written informed consent.
10. Study participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, dietary restrictions, and other study procedures.
11. No clinically significant abnormalities identified by medical history, physical examination, vital signs, ECG, and clinical laboratory tests in the opinion of the Investigator.

EXCLUSION: An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any prior use of the study test article, BIO 300 Oral Suspension, or the related test article BIO 300 Oral Powder.
2. Any known allergies to the study test article and its components (i.e., parabens)
3. Any clinically significant weight loss any time in prior 4 weeks at discretion of Investigator based on medical history interview.
4. Study participants with any of the following are not eligible;

   1. Previous history of QTc prolongation resulting from "known-risk" medications (www.Crediblemeds.org) that required discontinuation of that medication;
   2. Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age;
   3. Presence of left bundle branch block (LBBB);
   4. QTc with Fridericia's correction (QTcF) that is unmeasurable, or > 480 msec on screening or Day 1 pre-dose ECG. The average QTcF from the screening and Day 1 pre-dose ECG (completed in triplicate) must be ≤ 480 msec in order for the study participant to be eligible for the study. Based on the initial triplicate results, if in the opinion of the Investigator it is warranted, the screening or Day 1 pre-dose ECG can be repeated one time in triplicate to determine study participant eligibility.
5. Study participants with a history of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or atrial fibrillation) which is symptomatic or requires treatment (CTCAE Grade 3) or asymptomatic sustained ventricular tachycardia are not eligible.
6. Psychiatric conditions, social situations or substance abuse that precludes the ability of the study participant to cooperate with the requirements of the trial and protocol therapy at Investigator discretion.
7. Inability to refrain from alcohol consumption for 48 hours prior to day 1 and for the duration of the study or THC use from screening to day 1 and for the duration of the study. Illicit drugs must be avoided from screening through the duration of the study.
8. Positive results for Hep B surface antigen, Hep C antibody, or HIV 1/2 antibody at screening visit. Positive Hep C antibody test allowed if reflex test is negative.
9. Clinically significant immunodeficiency disorder in the opinion of the Investigator.
10. Pregnancy or women and men who are sexually active and not willing/able to use effective methods of contraception.
11. Participants who are actively breastfeeding are not eligible for this study.
12. Study participants that consume a soy-rich diet in the opinion of the Investigator such as participants that are vegan or vegetarian.
13. Any history of systemic infection requiring hospitalization, systemic antibiotics, or as judged clinically significant by the Investigator in the 3 months prior to day 1.
14. Any condition possibly affecting drug absorption (e.g., prior bariatric surgery, gastrectomy, intestinal resection). Participants who have undergone appendectomy or cholecystectomy are allowed so long as the surgery occurred more than 6 months prior to day 1.
15. Treatment with another investigational drug within 30 days or 5 half-lives (whichever is longer) proceeding Day 1 and during the duration of the study.
16. Positive drug screen or alcohol test at screening and day 1 predose. Positive THC screen allowed at screening but must be negative on day 1.
17. Blood donation of approximately 1 pint (500 ml) or more within 60 days of day 1; plasma donations within 14 days of day 1. Study participants must agree not to donate blood or plasma for the duration of the study and for 7 days following the end of study procedures.
18. Study participants must agree not to donate ova (eggs) or sperm for the duration of the study and for 7 days following the last dose of study drug.
19. Inability to swallow liquid medication.
20. History of sensitivity to heparin or heparin-induced thrombocytopenia.
21. Participants recruited for the food effect study that cannot consume the entire standardized high fat meal without substitutions.
22. Any chronic condition that requires daily medication
23. Considered by the Investigator to be unsuitable to participate in the study for any other reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Describe the overall adverse event profile of BIO 300 Oral Suspension in healthy volunteers following repeat dosing or single doses under fed and fasted conditions | Up to 7 days after the last dose
  Report the incidence and severity of BIO 300 Oral Suspension-related adverse events following 14 days of once daily administration and single doses administered under fed vs fasted conditions as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Describe the effects of multiple ascending doses of BIO 300 Oral Suspension on gene expression in the blood as assessed by RNA sequencing | From enrollment to the end of treatment at 14 days
  Assess changes in differential gene expression in the whole blood related to BIO 300 Oral Suspension after 1, 6 and 14 days of dosing.
Describe the effects of multiple ascending doses of BIO 300 Oral Suspension on protein expression in the blood as assessed by proximity extension assay | From enrollment to the end of treatment at 14 days
  Assess changes in protein expression in the blood serum related to BIO 300 Oral Suspension after 1, 6 and 14 days of dosing.
Identify serum metabolites of genistein after single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | From enrollment to 48 hours after the last dose
  Report the serum metabolites of genistein and their relative abundance after 1 or 14 days of dosing
Evaluate the potential for BIO 300 Oral Suspension to prolongate the corrected QT (QTc) interval following single and repeat doses | From enrollment to 24 hours dosing
  Change in QTc interval relative to baseline following a single dose of BIO 300 Oral Suspension administered under fasted conditions
Evaluate the potential for BIO 300 Oral Suspension to prolongate the corrected QT (QTc) interval following single and repeat doses | From enrollment to 24 hours after the first dose and the last dose
  Change in QTc interval relative to baseline following a single dose and 14 repeat doses of BIO 300 Oral Suspension
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the dose
  Report area under the serum concentration versus time curve (AUC) after 1 dose
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report area under the serum concentration versus time curve (AUC) after 6 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report area under the serum concentration versus time curve (AUC) after 14 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the dose
  Report peak serum concentration (Cmax) after 1 dose
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report peak serum concentration (Cmax) after 6 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report peak serum concentration (Cmax) after 14 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the dose
  Report time to peak serum concentration (Tmax) after 1 dose
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report time to peak serum concentration (Tmax) after 6 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report time to peak serum concentration (Tmax) after 14 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the dose
  Report half-life (T1/2) after 1 dose
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report half-life (T1/2) after 6 once daily doses
Establish the PK of single and repeat doses of BIO 300 Oral Suspension under fed or fasted conditions | 48 hours after the last dose
  Report half-life (T1/2) after 14 once daily doses

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, LLC, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning at the time of results publication with no end date

REFERENCES:
- See also: Sponsor's Company Website — https://www.humaneticscorp.com